CLINICAL TRIAL: NCT03993379
Title: A Phase 2, Open-Label, Multi-cohort Study of PD-L1 Probody Therapeutic CX-072 in Combination With Other Anticancer Therapy in Adults With Solid Tumors
Brief Title: PROCLAIM: CX-072-002: Study of PD-L1 Probody Therapeutic CX-072 in Combination With Other Anticancer Therapy in Adults With Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: CytomX Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTMX-M-072-002
Record Dates: First submitted 2019-05-14; First posted 2019-06-20 (Actual); Results first posted 2021-12-01 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor; Unresectable or Metastatic Melanoma
Keywords: Combination; ipilimumab; Cancer; checkpoint inhibitor; PD-L1; CTLA-4; PROCLAIM; PROCLAIM-CX-072; Relapsed; Refractory
MeSH Terms: conditions — Melanoma; Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12; Recurrence | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CX-072 in combination with anti-cancer therapy-front line (Experimental): histologically or cytologically confirmed solid tumor who have received no prior treatment
  Interventions: Drug: CX-072
- CX-072 in combination with ipilimumab (Experimental): histologically or cytologically confirmed Stage III (unresectable) or Stage IV melanoma who have experienced progressive disease or relapse following treatment with a PD-1/PD-L1 immune checkpoint inhibitor
  Interventions: Drug: CX-072; Drug: Ipilimumab
- CX-072 in combination with anti-cancer therapy-Progressed (Experimental): histologically or cytologically confirmed, advanced/unresectable or metastatic solid tumor that have experienced disease progression during or following treatment with platinum based therapy
  Interventions: Drug: CX-072
- CX-072 in combination with anti-cancer therapy-Neoadjuvant (Experimental): neo-adjuvant study in subjects with histologically confirmed solid tumor
  Interventions: Drug: CX-072

INTERVENTIONS:
Drug: CX-072 — CX-072 in combination with ipilimumab
Drug: Ipilimumab — CX-072 in combination with ipilimumab
  Arms: CX-072 in combination with ipilimumab

SUMMARY:
To obtain evidence of antitumor effect of CX-072 in combination with anticancer therapy in adult patients with solid tumor based upon overall response rate by Response Evaluation Criteria in Solid Tumors (RECIST)

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Measurable disease as defined by RECIST v1.1
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤1
4. Agree to provide tumor tissue and blood samples for biomarker assessment

Exclusion Criteria:

1. Treatment with cytotoxic chemotherapy, biologic agents, radiation, immunotherapy, or any investigational agent within 28 days prior to the first dose of study treatment.
2. Prior therapy with a chimeric antigen receptor T cell-containing regimen
3. History of active autoimmune disease(s) including but not limited to inflammatory bowel diseases, rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic sclerosis, systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies, type 1 insulin-dependent diabetes mellitus
4. History of myocarditis regardless of the cause
5. History of intolerance to prior checkpoint inhibitor therapy defined as the need to discontinue treatment due to an irAE
6. History of any syndrome or medical condition that required treatment with systemic steroids (≥10 mg daily prednisone equivalents) or immunosuppressive medications.
7. History of severe allergic or anaphylactic reactions to human mAb therapy or known hypersensitivity to any Probody therapeutic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-05-21 (Actual); Study Completion 2020-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Lu, MD, Study Director — CytomX Therapeutics
Locations (27):
- United States (14):
  - City of Hope National Medical Center, Duarte, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - Beacon Cancer Care, Coeur d'Alene, Idaho
  - University of Chicago, Chicago, Illinois
  - Norton Cancer Institute, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - NYC Cancer Institute, New York, New York
  - Columbia Medical Center, New York, New York
  - Oregon Health & Science Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Inova Dwight and March Schar Cancer Institute, Fairfax, Virginia
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Multicare Institute for Research and Innovation, Spokane, Washington
- Australia (2):
  - Sunshine Coast University Private Hospital, Sunshine Coast, Queensland
  - Ballarat Oncology and Haematology Services, Wendouree, Victoria
- Netherlands (2):
  - The Netherlands Cancer Institute, Amsterdam
  - University Medical Center Groningen, Groningen
- South Korea (4):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
- Spain (5):
  - ICO Hospitalet, Hospital Duran I Reynals, Barcelona
  - Hospital Clinic de Barcelona. Servicio Oncologia Medica, Barcelona
  - Hospital Universitario La Paz, Madrid
  - START- Madrid, Madrid
  - Clinica Universitaria de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was composed of 2 parts (Part A and Part B) and 4 cohorts (A1, A2, A3, B1).
Pre-assignment Details: Subjects who meet Inclusion / Exclusion criteria began the Screening Period within 30 days prior to the first dose of study treatment. Subjects for whom consent was provided underwent Screening Period assessments to determine eligibility for the study; assessments were to be performed within 30 days prior to the first dose of study treatment.
Groups:
- Cohort A1: CX-072 in Combination With Anti-cancer Therapy-front Line: Histologically or cytologically confirmed solid tumor who have received no prior treatment
  CX-072 in combination with ipilimumab
  Part A Dosing Regimen:
  * Combination treatment: 800 mg CX-072 + 3 mg/kg ipilimumab, q3w
  * Monotherapy treatment: 800 mg CX-072, q2w
- Cohort A2: CX-072 in Combination With Ipilimumab: Histologically or cytologically confirmed Stage III (unresectable) or Stage IV melanoma who have experienced progressive disease or relapse following treatment with a PD-1/PD-L1 immune checkpoint inhibitor
  CX-072 in combination with ipilimumab
  Part A Dosing Regimen:
  * Combination treatment: 800 mg CX-072 + 3 mg/kg ipilimumab, q3w
  * Monotherapy treatment: 800 mg CX-072, q2w
- Cohort A3: CX-072 in Combination With Anti-cancer Therapy-Progressed: Histologically or cytologically confirmed, advanced/unresectable or metastatic solid tumor that have experienced disease progression during or following treatment with platinum based therapy
  CX-072 in combination with ipilimumab
  Part A Dosing Regimen:
  * Combination treatment: 800 mg CX-072 + 3 mg/kg ipilimumab, q3w
  * Monotherapy treatment: 800 mg CX-072, q2w
- Cohort B1: CX-072 in Combination With Anti-cancer Therapy-Neoadjuvant: Neo-adjuvant study in subjects with histologically confirmed solid tumor
  CX-072 in combination with ipilimumab
  Part B Dosing Regimen:
  * Combination treatment: 800 mg CX-072 + 1 mg/kg ipilimumab, q3w
  * Monotherapy treatment: 800 mg CX-072, q2w
Period: Overall Study
Arm/Group | Cohort A1: CX-072 in Combination With Anti-cancer Therapy-front Line | Cohort A2: CX-072 in Combination With Ipilimumab | Cohort A3: CX-072 in Combination With Anti-cancer Therapy-Progressed | Cohort B1: CX-072 in Combination With Anti-cancer Therapy-Neoadjuvant
Started | 0 | 3 | 0 | 0
Completed | 0 (No subjects enrolled in this arm/group.) | 0 (Subjects did not complete due to early termination of the study due to business reasons.) | 0 (No subjects enrolled in this arm/group.) | 0 (No subjects enrolled in this arm/group.)
Not Completed | 0 | 3 | 0 | 0
Not completed — The study was terminated early due to business decision. | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Due to the early study termination, a statistical analysis plan was not generated. The statistical analyses per the study protocol were not performed due to insufficient sample size and the efficacy and pharmacokinetic analyses were not performed.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A1: CX-072 in Combination With Anti-cancer Therapy-front Line | Cohort A2: CX-072 in Combination With Ipilimumab | Cohort A3: CX-072 in Combination With Anti-cancer Therapy-Progressed | Cohort B1: CX-072 in Combination With Anti-cancer Therapy-Neoadjuvant | Total
Number analyzed (Participants) | 0 | 3 | 0 | 0 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 0 | 0 | 1
  >=65 years | 0 | 2 | 0 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 0 | 1
  Male | 0 | 2 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | 0 |  |  | 0
  Asian |  | 1 |  |  | 1
  Native Hawaiian or Other Pacific Islander |  | 0 |  |  | 0
  Black or African American |  | 0 |  |  | 0
  White |  | 2 |  |  | 2
  More than one race |  | 0 |  |  | 0
  Unknown or Not Reported |  | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  Netherlands |  | 0 |  |  | 0
  South Korea |  | 0 |  |  | 0
  United States |  | 3 |  |  | 3
  Australia |  | 0 |  |  | 0
  Spain |  | 0 |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate by RECIST v 1.1
Description: ORR by RECIST v1.1
Time Frame: 1 year
Population: All subjects who have at least one measurable lesion at baseline, receive at least 1 infusion of CX-072 DP and have at least 1 postbaseline RECIST 1.1 assessment, or who discontinue treatment/study due to disease progression by RECIST v 1.1.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: CX-072 in Combination With Anti-cancer Therapy-front Line | Cohort A2: CX-072 in Combination With Ipilimumab | Cohort A3: CX-072 in Combination With Anti-cancer Therapy-Progressed | Cohort B1: CX-072 in Combination With Anti-cancer Therapy-Neoadjuvant
Number analyzed (Participants) | 0 | 2 | 0 | 0
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0
  Partial Response (PR) | 0 | 0 | 0 | 0
  Stable Disease (SD) | 0 | 0 | 0 | 0
  Progressive Disease (PD) | 0 | 2 | 0 | 0

2. Secondary Outcome: The Percentage of Patients Experiencing Treatment Related Adverse Events
Description: Safety and Tolerability of CX-072 in Combination Therapy
Time Frame: 2 years
Population: All subjects who receive any amount of CX-072.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: CX-072 in Combination With Anti-cancer Therapy-front Line | Cohort A2: CX-072 in Combination With Ipilimumab | Cohort A3: CX-072 in Combination With Anti-cancer Therapy-Progressed | Cohort B1: CX-072 in Combination With Anti-cancer Therapy-Neoadjuvant
Number analyzed (Participants) | 0 | 3 | 0 | 0
Participants
  Gastrointestinal disorders - Diarrhea (treatment related): Experienced | 0 | 1 | 0 | 0
  Gastrointestinal disorders - Diarrhea (treatment related): Did not experience | 0 | 2 | 0 | 0
  Hepatobiliary Disorders - Immune-mediated Hepatitis (treatment related): Experienced | 0 | 2 | 0 | 0
  Hepatobiliary Disorders - Immune-mediated Hepatitis (treatment related): Did not experience | 0 | 1 | 0 | 0
  Gastrointestinal disorders - Vomitting (treatment related): Experienced | 0 | 1 | 0 | 0
  Gastrointestinal disorders - Vomitting (treatment related): Did not experience | 0 | 2 | 0 | 0
  Metabolism and nutrition disorders - Dehydration (treatment related): Experienced | 0 | 1 | 0 | 0
  Metabolism and nutrition disorders - Dehydration (treatment related): Did not experience | 0 | 2 | 0 | 0
  Skin and subcutaneous tissuedisorders - Rash Generalized (treatment related): Experienced | 0 | 1 | 0 | 0
  Skin and subcutaneous tissuedisorders - Rash Generalized (treatment related): Did not experience | 0 | 2 | 0 | 0
  Injury, poisoning and proceduralcomplications - Infusion Related Reaction: Experienced | 0 | 1 | 0 | 0
  Injury, poisoning and proceduralcomplications - Infusion Related Reaction: Did not experience | 0 | 2 | 0 | 0

3. Secondary Outcome: The Numbers of Patients Experiencing Anti-tumor Activity by irRECIST
Description: ORR by irRECIST
Time Frame: 2 years
Population: All subjects who have at least one measurable lesion at baseline, receive at least 1 infusion of CX-072 DP and have at least 1 postbaseline irRECIST assessment, or who discontinue treatment/study due to disease progression by irRECIST.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A1: CX-072 in Combination With Anti-cancer Therapy-front Line | Cohort A2: CX-072 in Combination With Ipilimumab | Cohort A3: CX-072 in Combination With Anti-cancer Therapy-Progressed | Cohort B1: CX-072 in Combination With Anti-cancer Therapy-Neoadjuvant
Number analyzed (Participants) | 0 | 2 | 0 | 0
Participants
  immune-related Complete Response (irCR) | 0 | 0 | 0 | 0
  immune-related Partial Response (irPR) | 0 | 0 | 0 | 0
  immune-related Stable Disease (irSD) | 0 | 0 | 0 | 0
  immune-related Progressive Disease (irPD) | 0 | 2 | 0 | 0
  no target disease identified at baseline and at follow-up (irNN) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The pre-specified AE reporting period spans from signing of the ICF to 30 days after the last dose. Monitoring continued for immune-related AEs, AEs ≥ Grade 3, and serious AEs (SAEs) up to 90 days following the last dose of the study drug. All AEs are reported from signing of the informed consent through study completion, an average of 4 months.
Description: All AEs are reported from signing of the informed consent through study completion, regardless of attribution/causality.
Arm/Group | Cohort A1: CX-072 in Combination With Anti-cancer Therapy-front Line | Cohort A2: CX-072 in Combination With Ipilimumab | Cohort A3: CX-072 in Combination With Anti-cancer Therapy-Progressed | Cohort B1: CX-072 in Combination With Anti-cancer Therapy-Neoadjuvant
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/3 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/3 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 3/3 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A1: CX-072 in Combination With Anti-cancer Therapy-front Line (N=0) | Cohort A2: CX-072 in Combination With Ipilimumab (N=3) | Cohort A3: CX-072 in Combination With Anti-cancer Therapy-Progressed (N=0) | Cohort B1: CX-072 in Combination With Anti-cancer Therapy-Neoadjuvant (N=0)
Immune-mediated Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A1: CX-072 in Combination With Anti-cancer Therapy-front Line (N=0) | Cohort A2: CX-072 in Combination With Ipilimumab (N=3) | Cohort A3: CX-072 in Combination With Anti-cancer Therapy-Progressed (N=0) | Cohort B1: CX-072 in Combination With Anti-cancer Therapy-Neoadjuvant (N=0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 1 (2) | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 1 (1) | 0 | 0
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 (1) | 0 | 0
Generalized Oedema (General disorders) | 0 | 1 (1) | 0 | 0
Oedema Peripheral (General disorders) | 0 | 1 (1) | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Vomitting (Gastrointestinal disorders) | 0 | 1 (1) | 0 | 0
Immune-mediated Hepatitis (Hepatobiliary disorders) | 0 | 2 (2) | 0 | 0
Rash Generalized (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 (2) | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 (1) | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 (1) | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0 | 0

LIMITATIONS AND CAVEATS:
Due to developmental strategic reasons and slow enrollment because of the COVID-19 pandemic, the study was terminated early. Three subjects were enrolled, all in Cohort A2. The last subject observation for this study was on 21 May 2020. Since the study terminated early, a statistical analysis plan was not generated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT03993379/Prot_SAP_001.pdf